CLINICAL TRIAL: NCT00004582
Title: A Phase II Study of ABT-378/Ritonavir and Efavirenz in Multiple Protease Inhibitor-Experienced Subjects
Brief Title: ABT-378/Ritonavir and Efavirenz in HIV-Infected Patients Who Have Taken More Than One Protease Inhibitor in the Past
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViRx (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 285E; M98-957
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-08

CONDITIONS: HIV Infections
Keywords: HIV Protease Inhibitors; Ritonavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; ABT 378; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; efavirenz

INTERVENTIONS:
Drug: Lopinavir/Ritonavir
Drug: Efavirenz

SUMMARY:
The purpose of this study is to see if ABT-378/ritonavir plus efavirenz is safe and effective in lowering the amount of HIV in the blood of patients who have been treated with more than 1 protease inhibitor (PI).

DETAILED DESCRIPTION:
All patients take ABT-378/ritonavir and efavirenz; there are no placebos in this study. Patients take study medications for 48 weeks, during which time there will be 15 study visits. There is a possibility of a study extension after 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a viral load (level of HIV in the blood) of at least 1,000 copies/ml.
* Have been receiving stable (no changes) anti-HIV treatment that includes at least 1 PI for at least 8 weeks prior to study entry.
* Have received more than 1 PI for at least 12 weeks each at some time in the past.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have had any active opportunistic (AIDS-related) infections within the past 30 days.
* Have ever received nonnucleoside reverse transcriptase inhibitors (NNRTIs), such as delavirdine, nevirapine, or efavirenz.
* Have received certain medications.
* Are pregnant or breast-feeding.
* Abuse alcohol or drugs.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- ViRx Inc, San Francisco, California, United States